CLINICAL TRIAL: NCT04258696
Title: Assessment of Lateral and Vertical Tissue Displacement Obtained by the Retraction Cord and Diode Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Abdelzaher Abdelhamid Omara, Lecturer assistant , Fixed Prosthodontics Department ,Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2019-09-30
Record Dates: First submitted 2019-11-01; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Endodontically-Treated Teeth; Spacing of Anterior Maxillary Teeth; Broken Teeth Injury With Complication
Keywords: Gingival retraction; Gingival displacement; Diode laser
MeSH Terms: conditions — Tooth, Nonvital | interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gingival retraction by ultrapak retraction cord (Active Comparator)
  Interventions: Device: ultrapak Knitted retraction cord
- Gingival retraction by diode laser (Experimental)
  Interventions: Device: diode laser

INTERVENTIONS:
Device: diode laser — using Ultrapak Knitted retraction cord as a gingival retraction method . using Wiser Cordless Dental Diode Laser from Doctor Smile Dental Laser By LAMBDA SpA Italy as a gingival retraction method.• The tip of diode laser, will be angled toward the soft tissue and away from the prepared tooth, will be passed along the gingival sulcus to remove the sulcular epithelium. Constant and steady short brushing strokes gently removed the lining of the sulcus in order to achieve a full 360-degree trough. The tip will be constantly cleaned with a gauze sponge wetted with hydrogen peroxide to remove debris and to eliminate potential bacterial contamination. sufﬁcient epithelium will be removed to place the impression material and visualize the ﬁnishing line. The tissue will be kept moist with water during the procedure then impression will be taken
  Arms: Gingival retraction by diode laser
Device: ultrapak Knitted retraction cord — using Ultrapak Knitted retraction cord as a gingival retraction method retraction cord will be applied for 8-10 mins then an impression will be taken , poured to obtain a cast and the die sectioned
  Arms: Gingival retraction by ultrapak retraction cord

SUMMARY:
In fixed prosthodontic treatment, deflection of gingival tissues for diagnosis or making an impression is one of the important phases. Gingival displacement is defined as "displacement of gingival tissues both in vertical and lateral dimensions". Lateral retraction displaces the tissues so that an adequate bulk of impression material can be interfaced with the prepared tooth. Vertical retraction exposes the uncut portion of the tooth apical to the finish line Conventional gingival retraction cord technique may injure the healthy epithelial lining and result in postoperative gingival recession The diode laser has been used for displacing gingiva to make a deﬁnitive impression. Rather than displacing gingival tissue, it removes the epithelial lining from the sulcus.

The aim of the Study is to compare between the Ultrapak retraction cord and diode laser regarding the amount of vertical and lateral retraction and patient comfort.

ELIGIBILITY:
Inclusion Criteria:

* Age range of the patients from 20-45 years old; able to read and sign the informed consent document, illiterate patient will be avoided.
* Patients able physically and psychologically to tolerate conventional restorative procedures.
* Patients with no active periodontal disease.
* Patients with thick gingival biotype.
* Patients with teeth problems indicated for full coverage restoration .
* Vital or non vital teeth.
* Good Oral hygiene.

Exclusion Criteria:

* Patients with poor oral hygiene.
* Patients with thin gingival biotype.
* Pregnant women.
* Unmotivated patients.
* Patients with gingival recession.
* Patients with psychiatric problems or unrealistic expectation .
* patient suffer from parafunctional habit .
* Smokers and heavy caffeine consumers.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-06-30 (Estimated); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Amount of lateral tissue displacement | through study completion,up to 24 weeks
  Measured using Stereomicroscope

SECONDARY OUTCOMES:
Amount of vertical tissue displacement | through study completion,up to 24 weeks
  Measured using Stereomicroscope

OTHER OUTCOMES:
Patient satisfaction | through study completion,up to 24 weeks
  Pain scale ( 0 - 5 ) 5 means maximum pain, worse outcome , 1 means low pain,better outcome
  o means no pain

CONTACTS AND LOCATIONS:
Locations (1):
- Alaa Abdelzaher Abdelhamid Omara, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided